CLINICAL TRIAL: NCT02802020
Title: Fully Covered Self Expanding Metal Stents (FCSEMS) for Pancreatic Duct Strictures in Patients With Chronic Pancreatitis
Brief Title: WallFlex Pancreatic Metal Stent for Pancreatic Duct Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7104
Record Dates: First submitted 2016-05-16; First posted 2016-06-16 (Estimated); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- WallFlex FCSEMS Recipients (Experimental): The WallFlex™ Pancreatic RX Fully Covered Soft Stent System consists of a flexible delivery system preloaded with a self-expanding pancreatic metal stent. Patients who meet all eligibility criteria will receive the WallFlex Pancreatic stent for up to 6 months stent indwell and 6 months follow-up after stent removal. A patient is considered "enrolled" after signing the study-specific Informed Consent Form (ICF). Patients who sign the ICF but subsequently do not meet one or more of the selection criteria will be considered screen failures and excluded from the study.
  Interventions: Device: Pancreatic fully-covered self-expanding metal stent (FCSEMS)

INTERVENTIONS:
Device: Pancreatic fully-covered self-expanding metal stent (FCSEMS) — The WallFlex™ Pancreatic RX Fully Covered Soft Stent System consists of a flexible delivery system preloaded with a self-expanding pancreatic metal stent.
  Other Names: WallFlex

SUMMARY:
To prospectively document the performance of a FCSEMS for treatment of pancreatic duct strictures in patients with painful chronic pancreatitis.

DETAILED DESCRIPTION:
This study is a prospective, single arm, pre-approval study. Treatment of up to 92 patients will take place at up to 15 clinical centers. Patient who meet all eligibility criteria will receive the WallFlex Pancreatic stent for up to 6 months stent indwell and 6 months follow-up after stent removal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to comply with study procedures and follow-up schedule and provide written informed consent to participate in study
* Chronic pancreatitis induced stricture of Cremer Type IV, namely distal dominant stricture with upstream ductal dilation.
* For patients with one prior plastic pancreatic stent: VAS Pain Score and Frequency of Pain sectors of the Izbicki pain scale at the time of placement of the plastic stent.
* Availability of narcotic dosage for at least one month prior to baseline visit for patients who do not have a prior plastic stent or availability for one month prior to placement of prior plastic stent, where applicable.
* VAS Pain Score of ≥ 20 before study stent placement for patients without a prior plastic pancreatic stent. VAS Pain Score of ≥ 20 before initial plastic pancreatic stent placement for patients with a prior plastic pancreatic stent indwelling for 90 days or less before study stent placement. VAS Pain Score is captured via Izbicki pain scale.
* Pain occurring weekly or more frequently (assessed by Frequency of Pain sector of the Izbicki pain scale) as reported before study stent placement for patients without a prior plastic pancreatic stent, or before placement of initial plastic pancreatic stent for patients with a prior plastic pancreatic stent indwelling for 90 days or less before study stent placement.
* Minimum 5 mm diameter of dilated duct immediately upstream of pancreatic duct stricture
* Prior clearance of pancreatic stones where needed

  * If pancreatic duct stone clearance prior to placement of the study stent includes ESWL, then a plastic pancreatic stent may be placed immediately after the ESWL procedure at the discretion of the Investigator, for example, if there is concern about stone fragments of stone sludge in side branches of the pancreatic duct, and may be left indwelling for 30-90 days.
  * If new pancreatic duct stones requiring ESWL have formed by the time of intended study stent placement, then the patient will not receive the study stent and be excluded from the study. Further treatment of the patient will be provided per standard of practice outside of the study. In case the study stent is not placed during the same session in which the plastic stent is removed, the pain score needs to be collected again prior to study stent placement.
* Prior endoscopic pancreatic sphincterotomy (EPS), historically or to be provided at time of SEMS placement as applicable.

Exclusion Criteria:

* Pancreatic or peri-ampullary cancer with or without pancreatic duct strictures caused by malignancy
* Biliary strictures caused by chronic pancreatitis that are symptomatic and/or in need of therapeutic intervention
* Perforated duct
* Ansa pancreatica
* Presence of pancreatic cysts suspected to be cystic tumor or requiring transmural drainage
* Duodenal/groove pancreatitis
* Autoimmune pancreatitis
* Pancreatic duct stenoses not located in the head of the pancreas
* Failed access during an attempted ERCP on a prior date at the investigational center
* Duration of indwell of one single plastic pancreatic stent or cumulative duration of consecutive single plastic pancreatic stents immediately prior to study stent placement exceeding 90 days
* History of prior single pancreatic plastic stent(s) followed by a stent-free period shorter than 1 year before enrollment into the study
* History of prior side-by-side multiple pancreatic plastic stents up to one year prior to enrollment
* History of prior pancreatic metal stent(s)
* Reported recent history of acute relapsing pancreatitis in the absence of chronic pancreatitis
* Patients for whom endoscopic techniques are contraindicated
* Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* Inability or refusal to comply with the follow-up schedule including patients living at such a distance from the investigational center that attending follow-up visits would be unusually difficult or burdensome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, MD, PhD, Principal Investigator — ULB Erasme Hospital
Locations (11):
- United States (6):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Indiana University Health Medical Center, Indianapolis, Indiana
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- ULB Erasme Hospital, Brussels, Belgium
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India
- Policlinico A. Gemelli, Rome, Italy
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherman S, Kozarek RA, Costamagna G, Reddy DN, Tarnasky P, Shah RJ, Slivka A, Fogel E, Watkins J, Delhaye M, Irani SS, Tringali A, Lakhtakia S, Kedia P, Edmundowicz S, Peetermans JA, Rousseau MJ, Deviere J; Pancreatic SEMS in Chronic Pancreatitis Study Group. Soft self-expandable metal stent to treat painful pancreatic duct strictures secondary to chronic pancreatitis: a prospective multicenter trial. Gastrointest Endosc. 2023 Mar;97(3):472-481.e3. doi: 10.1016/j.gie.2022.09.021. Epub 2022 Oct 5. PMID 36208796

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered "enrolled" after providing written informed consent. Participants who provided written informed consent but subsequently did not meet one or more of the selection criteria were considered screen failures and excluded from the study. Only participants who met all eligibility criteria were counted toward the enrollment ceiling and considered the primary analysis cohort.
Period: Overall Study
Arm/Group | WallFlex FCSEMS Recipients
Started | 67
Completed | 63
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 9
  India | 7
  Italy | 7
  United States | 44
Time Since CP Diagnosed [Mean (Standard Deviation); unit: years] — Population: The number of participants analyzed for time since CP diagnosis is lower than the number of baseline participants due to missing data or status unknown.
  years
    number analyzed (Participants) | 23
    (all) | 6.4 (6.4)
Weight [Mean (Standard Deviation); unit: kilograms] | 71.5 (18.4)
CP Etiology [Count of Participants; unit: Participants]
  Alcoholic | 33
  Hereditary | 3
  Gallstones | 1
  Smoking | 24
  Other | 8
  Unknown | 19
Current Alcohol Consumption [Count of Participants; unit: Participants] | 8
CP Calcific [Count of Participants; unit: Participants]
  Yes | 48
  No | 18
  Unknown | 1
Type of Calcification [Count of Participants; unit: Participants] — Population: Of the 67 baseline participants, 48 participants were reported to have calcific CP. As a result, only 48 participants were evaluated for type of calcification.
  Participants
    number analyzed (Participants) | 48
    Ductal | 20
    Parenchymal | 9
    Both | 19
Surgical Candidate [Count of Participants; unit: Participants]
  Yes | 46
  No | 12
  Unknown | 9
Smoking Status [Count of Participants; unit: Participants]
  Current | 36
  Previous | 17
  Never | 14
Narcotic Dose [Mean (Standard Deviation); unit: morphine milligram equivalents] — Population: The number of participants analyzed for narcotic dose is lower than the number of baseline participants due to missing data or status unknown.
  morphine milligram equivalents
    number analyzed (Participants) | 65
    (all) | 31.9 (52.3)
Time Since First Narcotic Medication [Mean (Standard Deviation); unit: years] — Population: The number of participants analyzed for time since first narcotic medication is lower than the number of baseline participants due to missing data or status unknown.
  years
    number analyzed (Participants) | 28
    (all) | 4.8 (7.3)
Steatorrhea [Count of Participants; unit: Participants] | 13
Diabetes Status [Count of Participants; unit: Participants]
  Insulin Dependent | 20
  Oral Medication | 5
Pancreas Divisum [Count of Participants; unit: Participants] | 18
Prior Pancreatic Sphincterotomy Performed [Count of Participants; unit: Participants] | 47
Prior Biliary or Pancreatic Sphincterotomy Performed [Count of Participants; unit: Participants] | 48
History of Pancreatic Duct Stones [Count of Participants; unit: Participants]
  Yes | 37
  Unknown | 4
Stone Clearance Procedures Performed [Count of Participants; unit: Participants] — Population: Of the 67 baseline participants, 31 participants were reported to have stone clearance procedures performed. As a result, only 31 participants were evaluated for type of stone clearance procedure(s) performed.
  Participants
    ESWL: number analyzed (Participants) | 31
    ESWL | 16
    Balloon: number analyzed (Participants) | 31
    Balloon | 20
    Basket: number analyzed (Participants) | 31
    Basket | 5
    Other: number analyzed (Participants) | 31
    Other | 1
Current Pancreatic Stones [Count of Participants; unit: Participants] | 42
Largest Stone [Mean (Standard Deviation); unit: millimeter] — Population: Of the 67 baseline participants, 42 participants were reported to have current pancreatic stones. Only 40 participants were evaluated for largest stone size. The number of participants analyzed for largest stone size is lower than the number of participants with current pancreatic stones due to missing data or status unknown.
  millimeter
    number analyzed (Participants) | 40
    (all) | 6.2 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain Reduction
Description: The self-reported pain score (0-100) was the mean of the Visual Analogue Scale (VAS) and Izbicki Frequency of Pain subscore (sum treated as a continuous variable).The primary efficacy endpoint was the proportion of patients who had complete (pain score ≤ 10) or partial (pain score ˃ 10 but reduced at least 50% compared to pain as baseline) pain relief by 6 months after FCSEMS removal or observation of CDM or partial stent migration. Primary efficacy endpoint failure included any of the following: 1) no pain relief, 2) complete or partial pain relief in the setting of a 50% higher average daily narcotic dose compared to the patient's daily average narcotic dose in the month prior to baseline and at 6 months post-stent removal/observation of CDM, 3) stent migration in setting of recurring pain (VAS Pain Score of ≥ 20), 4) restenting in the setting of recurring pain.
Time Frame: Baseline to 6 months post-stent removal or 6 months post-observation of complete or partial stent migration
Population: There were 67 participants who enrolled in the study and had attempted FCSEMS placement. Of the 67 participants with attempted FCSEMS placement, 21 were excluded because they were not eligible for the primary efficacy endpoint analysis (i.e., 16 had insufficient pain, 2 died, and 3 were lost to follow-up). As a result, 46 participants were eligible for the primary efficacy endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 46
Participants | 12
Statistical Analysis 1: Comparison: WallFlex FCSEMS Recipients; We hypothesized that "pain reduction" (as defined in Study endpoints above) would be achieved in a performance goal of at least 53% of patients receiving the study SEMS. Assuming an observed pain reduction rate of 75% and using an exact test with a one-sided alpha of 0.025, 43 patients were required to obtain power of at least 80%; Test type: Superiority; p = 0.999, Fisher Exact

2. Primary Outcome: Rate of Related SAEs From WallFlex Pancreatic Stent Placement to End of Study
Description: The primary safety endpoint was the rate of serious adverse events (SAEs) related to the FCSEMS or study procedures from FCSEMS placement to end of study follow-up. Pain thought to be caused by FCSEMS pancreatic stent expansion was reported but did not count towards the endpoint if all three of the following conditions applied:
  1. Pain managed by medication, with the exception of injectable narcotic use for more than 24 hours.
  2. Pain not causing pancreatic FCSEMS removal.
  3. Pain resolved by 72 hours after pancreatic FCSEMS placement.
Time Frame: Baseline to 6 months post-stent removal or 6 months post-observation of complete or partial stent migration
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 67
Participants | 21
Statistical Analysis 1: Comparison: WallFlex FCSEMS Recipients; Test type: Superiority — we hypothesized that the proportion of patients reporting one or more related SAE(s) would be below a performance goal of 32%. Assuming an observed SAE rate of 15% and using an exact test with one-sided alpha of 0.025, 57 patients were required to obtain power of at least 80%; p = 0.513, Fisher Exact

3. Secondary Outcome: Stent Placement Success
Description: Satisfactory position is defined as the stent being across the stricture, without visible occluding impaction at the genu of the pancreatic duct and with distal end of the stent visible in the duodenum.
Time Frame: Assessed upon study stent placement. This endpoint is assessed at the Study Stent Placement visit (Day 0).
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 67
Participants | 65

4. Secondary Outcome: Endoscopic Stent Removal Success
Description: Endoscopic stent removal success is defined as ability to remove stent endoscopically (forceps, snare) without serious stent removal-related adverse events.
Time Frame: Assessed at study stent removal or observation of complete or partial stent migration. This is endpoint is assessed through the Month 6 Study Stent Removal visit.
Population: There were 67 participants who enrolled in the study and had attempted FCSEMS placement. Technical success (i.e., successful stent placement) was achieved in 65 of the 67 participants with attempted FCSEMS placement. As a result, 65 participants were evaluated for the endoscopic stent removal success endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 65
Participants | 63

5. Secondary Outcome: Stent Migration Rate
Description: Stent migration is the change in location of a stent from its originally placed location. In this study, pancreatic stent migration was noted as partial or complete and either proximal (i.e., into the pancreas) or distal (i.e., out of the pancreas).
Time Frame: Study stent placement through 6 months post-stent removal or 6 months post-observation of complete or partial stent migration
Population: There were 67 participants who enrolled in the study and had attempted FCSEMS placement. Technical success (i.e., successful stent placement) was achieved in 65 of the 67 participants with attempted FCSEMS placement. As a result, 65 participants were evaluated for the stent migration endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 65
Participants | 31

6. Secondary Outcome: Restenting Rate
Description: Restenting is the placement of a non-study stent due to no improvement in clinical status and associated persistence of stricture following removal or complete distal migration of the study stent.
Time Frame: Study stent removal or observation of study stent migration through 6 months post-stent removal or 6 months post-observation of complete or partial stent migration
Population: There were 67 participants who enrolled in the study and had attempted FCSEMS placement. Technical success (i.e., successful stent placement) was achieved in 65 of the 67 participants with attempted FCSEMS placement. As a result, 65 participants were evaluated for the restenting rate endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 65
Participants | 11

7. Secondary Outcome: Secondary Stricture Rate
Description: A secondary stricture is a ductal narrowing located at the intraductal edge of the study stent.
Time Frame: as for outcome 5
Population: There were 67 participants who enrolled in the study and had attempted FCSEMS placement. Technical success (i.e., successful stent placement) was achieved in 65 of the 67 participants with attempted FCSEMS placement. As a result, 65 participants were evaluated for the secondary stricture rate endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex FCSEMS Recipients
Number analyzed (Participants) | 65
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from beginning of study participation until end of study, or approximately 12-15 months.
Arm/Group | WallFlex FCSEMS Recipients
All-Cause Mortality (participants affected / at risk) | 2/67
Serious Adverse Events (participants affected / at risk) | 21/67
Other Adverse Events (participants affected / at risk) | 20/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex FCSEMS Recipients (N=67)
Pain (Gastrointestinal disorders) | 10 (12)
Post-ERCP pancreatitis (Gastrointestinal disorders) | 8 (8)
Chronic pancreatitis exacerbation (Gastrointestinal disorders) | 3 (3)
Duodenal ulceration (Gastrointestinal disorders) | 1 (1)
Elevated liver function tests (Investigations) | 1 (1)
Ampullary occlusion of the bile duct (Hepatobiliary disorders) | 1 (1)
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 (1)
Portal vein and SMV thrombosis (Vascular disorders) | 1 (1)
Fatal multiorgan failure from sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex FCSEMS Recipients (N=67)
Abdominal Pain (Gastrointestinal disorders) | 18 (21)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Cholangitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02802020/Prot_SAP_000.pdf